CLINICAL TRIAL: NCT00425542
Title: Outpatient Treatment of Low-risk Patients With Pulmonary Embolism: a Randomized-controlled Trial
Brief Title: Safety Study of Outpatient Treatment for Pulmonary Embolism
Acronym: OTPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: Swiss National Science Foundation (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Drahomir Aujesky, MD, MSc, University of Lausanne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 3200B0-112165; 1R01HL085565-01A2 (NIH); NCT00974207 (obsolete NCT alias)
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2009-10

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary embolism; Outpatient care; Prognosis
MeSH Terms: conditions — Pulmonary Embolism | interventions — Ambulatory Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Outpatient treatment (Experimental)
  Interventions: Other: Outpatient care (vs traditional inpatient care)
- Inpatient care (No Intervention)

INTERVENTIONS:
Other: Outpatient care (vs traditional inpatient care) — Patients randomized to the outpatient arm are discharged from the emergency department within 24 hours after randomization. Patients randomized to the inpatient arm are admitted to the hospital and are discharged based on the decision of the managing physician at the hospital.
  Other Names: Ambulatory care
  Arms: Outpatient treatment

SUMMARY:
The purpose of this randomized clinical trial is to determine whether outpatient treatment is as effective and safe as inpatient treatment among low-risk patients with pulmonary embolism.

DETAILED DESCRIPTION:
Pulmonary embolism (PE) is a worldwide health problem, with an estimated incidence of up to 69 cases per 100,000 persons annually. In the U.S., 101,000 patients were hospitalized with a primary diagnosis of PE in 2002, resulting in direct medical costs of $720 million. There is growing evidence that outpatient treatment with low-molecular-weight heparin (LMWH) is an effective and safe option for up to 50% of patients with non-massive PE. Despite this evidence, outpatient treatment of PE is uncommon because (1) explicit criteria that identify patients who are at low-risk of adverse medical outcomes have not been available, and (2) randomized trials demonstrating the effectiveness and safety of outpatient treatment have not been performed. We developed a clinical prognostic model that accurately identifies patients with PE who are at low-risk for short-term mortality, symptomatic recurrent venous thromboembolism (VTE), and major bleeding. This model provides clinicians an easily applied, explicit risk stratification tool for patients with PE, addressing a key barrier to outpatient treatment. The broad objective of this clinical trial is to address the other major barrier to outpatient treatment of low-risk patients with non-massive PE, the effectiveness and safety of outpatient management. We will randomize low-risk patients (identified using our prognostic model) with PE from hospital emergency departments to receive outpatient or inpatient treatment with LMWH for ≥5 days, followed by oral anticoagulation. The specific aims of the project are to compare (1) the frequency of recurrent VTE, (2) the frequency of major bleeding and all-cause mortality, and (3) medical resource utilization and patient satisfaction with care among patients randomized to receive outpatient or inpatient treatment with LMWH. The primary study outcome will be the rate of symptomatic recurrent VTE at 3 months after randomization. The secondary outcomes will be the rate of major bleeding and all-cause mortality. The ancillary outcomes will be medical resource utilization and patient satisfaction with care. The hypotheses guiding this trial are that outpatient treatment with LMWH is as effective and safe as inpatient treatment with LMWH, and is also associated with reduced medical resource utilization and increase patient satisfaction with care. This study is innovative because it translates a validated prognostic model into clinical practice and represents the first direct comparison of outpatient versus inpatient treatment of low-risk patients with PE. Successful completion of this project will provide a strong scientific basis for treating low-risk patients with PE in the outpatient setting. Outpatient management of low-risk patients with PE is likely to improve quality and efficiency of care by reducing resource utilization and increasing patient satisfaction with care. Our findings will have importance to physicians, hospitals, and policy-makers who are committed to optimizing patient safety and providing high-quality, cost-effective care.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* objectively confirmed diagnosis of pulmonary embolism
* patients at low-risk (Pulmonary Embolism Severity Index score <=85)

Exclusion Criteria:

* patients at high-risk (Pulmonary Embolism Severity Index score >85)
* presence of hypoxemia (arterial SO2 <90% measured by pulse oximetry or an paO2 on room air of <60 mm Hg measured by blood gas analysis)
* systolic blood pressure of <100 mm Hg
* chest pain necessitating parenteral opioid administration
* active bleeding or at high-risk of major bleeding (stroke during the preceding 10 days, gastrointestinal bleeding during the preceding 14 days, or platelets <75,000 per mm3)
* renal failure (creatinine clearance of <30 ml/minute based on the Cockcroft-Gault formula)
* body mass >150 kg
* history of HIT or allergy to heparins
* therapeutic oral anticoagulation (INR ≥2)at the time of pulmonary embolism diagnosis
* potential barriers to treatment adherence or follow-up (alcoholism, illicit current or recent drug use, psychosis, dementia, homelessness, lack of telephone access, transportation time to nearest ED >45 minutes)
* known pregnancy
* imprisonment
* diagnosis of pulmonary embolism >23 hours ago
* refusal or inability to provide informed consent
* prior enrollment in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2007-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Recurrent, symptomatic venous thromboembolism (deep vein thrombosis or pulmonary embolism) | within 3 months of randomization

SECONDARY OUTCOMES:
Major bleeding | within 3 months of randomization
All-cause mortality | within 3 months of randomization
Patient satisfaction with care | within 2 weeks of randomization
Medical resource utilization | within 3 months of randomization

CONTACTS AND LOCATIONS:
Overall Officials: Drahomir Aujesky, MD, MSc, Principal Investigator — University of Lausanne, Switzerland; Donald M Yealy, MD, Principal Investigator — University of Pittsburgh
Locations (19):
- United States (3):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Carolinas Medical Center, Charlotte, North Carolina
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
- Belgium (2):
  - University Hospital Saint-Luc, Université Catholique de Louvain, Brussels
  - University of Leuven, Leuven
- France (10):
  - University of Angers, Angers
  - University of Argenteuil, Argenteuil
  - University of Boulogne, Boulogne
  - University Hospital of Brest, Brest
  - University of Clermont-Ferrand, Clermont-Ferrand
  - University of Dijon, Dijon
  - University of Nantes, Nantes
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Henri Mondor, Créteil, Paris
  - Thiers, Thiers
- Switzerland (4):
  - Kantonsspital Baden, Baden
  - University of Geneva, Geneva
  - University Hospital of Lausanne, Lausanne
  - Kantonsspital St. Gallen, Sankt Gallen

REFERENCES:
- [Background] Aujesky D, Obrosky DS, Stone RA, Auble TE, Perrier A, Cornuz J, Roy PM, Fine MJ. Derivation and validation of a prognostic model for pulmonary embolism. Am J Respir Crit Care Med. 2005 Oct 15;172(8):1041-6. doi: 10.1164/rccm.200506-862OC. Epub 2005 Jul 14. PMID 16020800
- [Background] Aujesky D, Roy PM, Le Manach CP, Verschuren F, Meyer G, Obrosky DS, Stone RA, Cornuz J, Fine MJ. Validation of a model to predict adverse outcomes in patients with pulmonary embolism. Eur Heart J. 2006 Feb;27(4):476-81. doi: 10.1093/eurheartj/ehi588. Epub 2005 Oct 5. PMID 16207738
- [Derived] Aujesky D, Roy PM, Verschuren F, Righini M, Osterwalder J, Egloff M, Renaud B, Verhamme P, Stone RA, Legall C, Sanchez O, Pugh NA, N'gako A, Cornuz J, Hugli O, Beer HJ, Perrier A, Fine MJ, Yealy DM. Outpatient versus inpatient treatment for patients with acute pulmonary embolism: an international, open-label, randomised, non-inferiority trial. Lancet. 2011 Jul 2;378(9785):41-8. doi: 10.1016/S0140-6736(11)60824-6. Epub 2011 Jun 22. PMID 21703676